CLINICAL TRIAL: NCT05876091
Title: Effects of Tobacco Flavoring and Liquid Composition on Vaping Topography
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of grant
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I 3234822; U54CA228110 (NIH)
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Tobacco-Related Carcinoma
MeSH Terms: interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vaping - (Experimental): Description The order of directed and ad libitum bouts are randomized within participants at each session.
  SESSION 1: Participants puff their own brand liquid on study.
  SESSIONS 2-5: Participants puff 1 of 4 randomly assigned tobacco flavor formulations at each visit on study.
  SESSIONS 6-7: Participants puff 1 of 2 randomly assigned nicotine formulations at each visit on study.
  Participants also undergo collection of saliva samples and optionally undergo collection of oral cell and oral rinse samples throughout study.
  Interventions: Other: Vaping; Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Other: Vaping — Undergo vape puffing regimen
  Other Names: Vape, Vaping
Procedure: Biospecimen Collection — Undergo collection of saliva samples and oral cell samples
  Other Names: Biological Sample Collection
Other: Questionnaire Administration — Administer Quesitonnaire

SUMMARY:
This clinical trial tests the effect of tobacco flavor and liquid composition on the way a person puffs on a vape (topography). In general, tobacco products are designed with sensory factors in mind, such as flavor, to increase the appeal. Flavors and the composition of nicotine, either made in a lab (synthetic) or from tobacco, may create positive sensory effects, such as look, feel and taste, and influence smoking behavior and willingness to try different types of cigarettes. Understanding how nicotine vaping products are used is important in assessing individual and population level health risks. Vape flavors and synthetic nicotine may be related to harmful effects on health from vaping and may impact the appeal, risk beliefs and vaping topography.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

* Examine the influence of tobacco flavoring composition on vaping topography.
* Examine the influence of synthetic versus (vs.) tobacco derived nicotine on vaping topography.

SECONDARY OBJECTIVE:

* Examine the influence of tobacco flavoring composition on vaping topography.
* Examine the influence of synthetic versus (vs.) tobacco derived nicotine on vaping topography.

OUTLINE:

The order of directed and ad libitum bouts are randomized within participants at each session.

SESSION 1: Participants puff their own brand liquid on study.

SESSIONS 2-5: Participants puff 1 of 4 randomly assigned tobacco flavor formulations at each visit on study.

SESSIONS 6-7: Participants puff 1 of 2 randomly assigned nicotine formulations at each visit on study.

Participants also undergo collection of saliva samples and optionally undergo collection of oral cell and oral rinse samples throughout study.

ELIGIBILITY:
Inclusion Criteria:

* Current daily vapers of products containing nicotine
* No daily concurrent use of other tobacco products
* Self-reported general good health
* Women of child bearing potential must be willing to provide a urine sample and test negative prior to receiving any study-related products/procedures
* Ability to speak, read, and write in English
* Participant must understand the investigational nature of this study and sign an independent ethics committee/institutional review board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Allergies - active untreated seasonal allergies that would interfere with smell or taste procedures
* Self-reported taste or smell deficits
* Pregnant or nursing female participants
* Medications known to interfere with taste/smell (i.e., certain nasal sprays, nasal antihistamines, decongestants, antibiotics, medications containing zinc)
* Unwilling to use open system vaping device in laboratory setting
* Positive diagnosis of human coronavirus 2019 infection (COVID-19) within 10 days prior to start of study intervention
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive the study intervention

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard O'Connor, Principal Investigator — Roswell Park
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study Population: SESSION 1: Participants puff their own brand liquid on study.
  SESSIONS 2-5: Participants puff 1 of 4 randomly assigned tobacco flavor formulations at each visit on study.
  SESSIONS 6-7: Participants puff 1 of 2 randomly assigned nicotine formulations at each visit on study.
Period: Session 1: Own Brand Topography
Arm/Group | Overall Study Population
Started | 18
Own Brand Directed Vaping | 18
Own Brand Ad Lib Vaping | 18
Completed | 18
Not Completed | 0
Period: Sessions 2-5: Tobacco Flavors
Arm/Group | Overall Study Population
Started | 18
Cowboy Liquid Ad Lib | 17
Cowboy Liquid Directed | 17
RY4 Liquid Ad Lib | 17
RY4 Liquid Directed | 17
Red Oak Liquid Ad Lib | 17
Red Oak Liquid Directed | 17
Unflavored Liquid Ad Lib | 17
Unflavored Liquid Directed | 17
Completed | 17
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Sessions 6-7: Nicotine Formulations
Arm/Group | Overall Study Population
Started | 17
Synthetic Liquid Ad Lib | 17
Synthetic Liquid Directed | 17
Tobacco Derived Liquid Ad Lib | 17
Tobacco Derived Liquid Directed | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Prospective participants completed 6-n-propylthiouracil (PROP), and sodium benzoate tasting, commonly used indicators linked to individual differences in sensory perception, using manufactured, pre-calibrated calibrated strips.
Groups:
- Vaping -: Description The order of directed and ad libitum bouts are randomized within participants at each session.
  SESSION 1: Participants puff their own brand liquid on study.
  SESSIONS 2-5: Participants puff 1 of 4 randomly assigned tobacco flavor formulations at each visit on study.
  SESSIONS 6-7: Participants puff 1 of 2 randomly assigned nicotine formulations at each visit on study.
  Participants also undergo collection of saliva samples and optionally undergo collection of oral cell and oral rinse samples throughout study.
  Vaping: Undergo vape puffing regimen
  Biospecimen Collection: Undergo collection of saliva samples and oral cell samples
  Questionnaire Administration: Administer Quesitonnaire
Arm/Group | Vaping -
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 7
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Puff Topography: Puff Count
Description: Measure of vaping topography counting total number of puffs.
Time Frame: Single Session, Approximately 2 hours in duration
Measure: Mean (Standard Error); unit: Number of Puffs
Groups:
- Session 1: Own Brand Puff Count Ad Lib: Mean ad lib puff count: Own Brand
- Session 1: Own Brand Puff Count Directed: Mean directed puff count: Own Brand
- Sessions 2-5: Cowboy Vaping Liquid Puff Count Ad Lib: Mean ad lib puff count: Cowboy vaping liquid
- Sessions 2-5: Cowboy Vaping Liquid Puff Count Directed: Mean directed puff count: Cowboy vaping liquid
- Sessions 2-5: RY4 Double Vaping Liquid Puff Count Ad Lib: Mean ad lib puff count: RY4 Double Vaping Liquid
- Sessions 2-5: RY4 Double Vaping Liquid Puff Count Directed: Mean directed puff count: RY4 Double vaping liquid
- Sessions 2-5: Unflavored Vaping Liquid Puff Count Ad Lib: Mean ad lib puff count: Unflavored vaping liquid
- Sessions 2-5: Unflavored Vaping Liquid Puff Count Directed: Mean directed puff count: Unflavored vaping liquid
- Sessions 2-5: Red Oak Vaping Liquid Puff Count Ad Lib: Mean ad lib puff count: Red Oak vaping liquid
- Sessions 2-5: Red Oak Vaping Liquid Puff Count Directed: Mean directed puff count: Red Oak vaping liquid
- Session 6-7: Synthetic Nicotine Liquid Puff Count Ad Lib: Mean ad lib puff count: Synthetic vaping liquid
- Session 6-7: Synthetic Nicotine Liquid Puff Count Directed: Mean directed ad lib puff count: Synthetic vaping liquid
- Session 6-7: Tobacco Derived Liquid Puff Count Ad Lib: Mean ad lib puff count: Tobacco Derived vaping liquid
- Session 6-7: Tobacco Derived Liquid Puff Count Directed: Mean directed puff count: Tobacco Derived vaping liquid
Arm/Group | Session 1: Own Brand Puff Count Ad Lib | Session 1: Own Brand Puff Count Directed | Sessions 2-5: Cowboy Vaping Liquid Puff Count Ad Lib | Sessions 2-5: Cowboy Vaping Liquid Puff Count Directed | Sessions 2-5: RY4 Double Vaping Liquid Puff Count Ad Lib | Sessions 2-5: RY4 Double Vaping Liquid Puff Count Directed | Sessions 2-5: Unflavored Vaping Liquid Puff Count Ad Lib | Sessions 2-5: Unflavored Vaping Liquid Puff Count Directed | Sessions 2-5: Red Oak Vaping Liquid Puff Count Ad Lib | Sessions 2-5: Red Oak Vaping Liquid Puff Count Directed | Session 6-7: Synthetic Nicotine Liquid Puff Count Ad Lib | Session 6-7: Synthetic Nicotine Liquid Puff Count Directed | Session 6-7: Tobacco Derived Liquid Puff Count Ad Lib | Session 6-7: Tobacco Derived Liquid Puff Count Directed
Number analyzed (Participants) | 18 | 18 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17
Number of Puffs | 13.9 (2.3) | 6.4 (0.8) | 13.2 (2.2) | 5.8 (0.8) | 15.4 (3.1) | 5.9 (0.9) | 13.2 (2.2) | 5.8 (0.9) | 13.0 (2.2) | 6.3 (1.2) | 14.3 (2.4) | 7.1 (0.9) | 13.4 (1.8) | 7.0 (0.9)

2. Primary Outcome: Puff Topography: Puff Duration (in Seconds)
Description: Measure of vaping topography counting duration of puffs in seconds.
Time Frame: Single Session, Approximately 2 hours in duration
Measure: Mean (Standard Error); unit: Mean Duration of Puffs (in seconds)
Groups:
- Session 1: Own Brand Puff Duration Ad Lib: Mean ad lib puff duration: Own Brand
- Session 1: Own Brand Puff Duration Directed: Mean directed puff duration: Own Brand
- Sessions 2-5: Cowboy Vaping Liquid Puff Duration Ad Lib: Mean ad lib puff duration: Cowboy vaping liquid
- Session 6-7: Synthetic Nicotine Liquid Puff Duration Ad Lib: Mean ad lib puff duration: Synthetic vaping liquid
- Session 6-7: Synthetic Nicotine Liquid Puff Duration Directed: Mean directed ad lib puff duration: Synthetic vaping liquid
- Session 6-7: Tobacco Derived Liquid Puff Duration Ad Lib: Mean ad lib puff duration: Tobacco Derived vaping liquid
- Session 6-7: Tobacco Derived Liquid Puff Duration Directed: Mean directed puff duration: Tobacco Derived vaping liquid
Arm/Group | Session 1: Own Brand Puff Duration Ad Lib | Session 1: Own Brand Puff Duration Directed | Sessions 2-5: Cowboy Vaping Liquid Puff Duration Ad Lib | Sessions 2-5: Cowboy Vaping Liquid Puff Count Directed | Sessions 2-5: RY4 Double Vaping Liquid Puff Count Ad Lib | Sessions 2-5: RY4 Double Vaping Liquid Puff Count Directed | Sessions 2-5: Unflavored Vaping Liquid Puff Count Ad Lib | Sessions 2-5: Unflavored Vaping Liquid Puff Count Directed | Sessions 2-5: Red Oak Vaping Liquid Puff Count Ad Lib | Sessions 2-5: Red Oak Vaping Liquid Puff Count Directed | Session 6-7: Synthetic Nicotine Liquid Puff Duration Ad Lib | Session 6-7: Synthetic Nicotine Liquid Puff Duration Directed | Session 6-7: Tobacco Derived Liquid Puff Duration Ad Lib | Session 6-7: Tobacco Derived Liquid Puff Duration Directed
Number analyzed (Participants) | 18 | 18 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17
Mean Duration of Puffs (in seconds) | 2.2 (0.3) | 3.5 (0.3) | 2.3 (0.3) | 3.1 (0.3) | 2.5 (0.4) | 3.0 (0.3) | 2.3 (0.3) | 3.2 (0.3) | 2.1 (0.2) | 2.9 (0.3) | 2.4 (0.4) | 3.0 (0.3) | 2.2 (0.3) | 2.9 (0.3)

3. Primary Outcome: Puff Topography: Inter Puff Interval (IPI)
Description: Measure of vaping topography counting the interval between puffs in seconds.
Time Frame: Single Session, Approximately 2 hours in duration
Measure: Mean (Standard Error); unit: Mean number of seconds between puffs
Groups:
- Session 1: Own Brand Inter Puff Interval Ad Lib: Mean ad lib inter puff interval: Own Brand
- Session 1: Own Brand Inter Puff Interval Directed: Mean directed inter puff interval: Own Brand
- Sessions 2-5: Cowboy Vaping Inter Puff Interval Ad Lib: Mean ad lib inter puff interval: Cowboy vaping liquid
- Sessions 2-5: Cowboy Vaping Liquid Inter Puff Interval Directed: Mean directed inter puff interval: Cowboy vaping liquid
- Sessions 2-5: RY4 Double Vaping Liquid Inter Puff Interval Ad Lib: Mean ad lib inter puff interval: RY4 Double Vaping Liquid
- Sessions 2-5: RY4 Double Vaping Liquid Inter Puff Interval Directed: Mean directed inter puff interval: RY4 Double vaping liquid
- Sessions 2-5: Unflavored Vaping Liquid Inter Puff Interval Ad Lib: Mean ad lib inter puff interval: Unflavored vaping liquid
- Sessions 2-5: Unflavored Vaping Liquid Inter Puff Interval Directed: Mean directed inter puff interval: Unflavored vaping liquid
- Sessions 2-5: Red Oak Vaping Liquid Inter Puff Interval Ad Lib: Mean ad lib inter puff interval: Red Oak vaping liquid
- Sessions 2-5: Red Oak Vaping Liquid Inter Puff Interval Directed: Mean directed inter puff interval: Red Oak vaping liquid
- Session 6-7: Synthetic Nicotine Liquid Inter Puff Interval Ad Lib: Mean ad lib inter puff interval: Synthetic vaping liquid
- Session 6-7: Synthetic Nicotine Liquid Inter Puff Interval Directed: Mean directed ad lib inter puff interval: Synthetic vaping liquid
- Session 6-7: Tobacco Derived Liquid Inter Puff Interval Ad Lib: Mean ad lib inter puff interval: Tobacco Derived vaping liquid
- Session 6-7: Tobacco Derived Liquid Inter Puff Interval Directed: Mean directed inter puff interval: Tobacco Derived vaping liquid
Arm/Group | Session 1: Own Brand Inter Puff Interval Ad Lib | Session 1: Own Brand Inter Puff Interval Directed | Sessions 2-5: Cowboy Vaping Inter Puff Interval Ad Lib | Sessions 2-5: Cowboy Vaping Liquid Inter Puff Interval Directed | Sessions 2-5: RY4 Double Vaping Liquid Inter Puff Interval Ad Lib | Sessions 2-5: RY4 Double Vaping Liquid Inter Puff Interval Directed | Sessions 2-5: Unflavored Vaping Liquid Inter Puff Interval Ad Lib | Sessions 2-5: Unflavored Vaping Liquid Inter Puff Interval Directed | Sessions 2-5: Red Oak Vaping Liquid Inter Puff Interval Ad Lib | Sessions 2-5: Red Oak Vaping Liquid Inter Puff Interval Directed | Session 6-7: Synthetic Nicotine Liquid Inter Puff Interval Ad Lib | Session 6-7: Synthetic Nicotine Liquid Inter Puff Interval Directed | Session 6-7: Tobacco Derived Liquid Inter Puff Interval Ad Lib | Session 6-7: Tobacco Derived Liquid Inter Puff Interval Directed
Number analyzed (Participants) | 18 | 18 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17
Mean number of seconds between puffs | 82.2 (14.0) | 55.2 (6.1) | 61.4 (10.7) | 58.0 (4.2) | 71.6 (10.3) | 54.2 (3.6) | 71.6 (8.7) | 56.7 (4.0) | 55.1 (8.1) | 60.6 (5.4) | 84.6 (12.0) | 59.3 (4.1) | 78.7 (11.0) | 56.6 (3.5)

4. Primary Outcome: Puff Topography: Puff Volume
Description: Measure of vaping topography measuring the volume per puff in ml.
Time Frame: Single Session, Approximately 2 hours in duration
Measure: Mean (Standard Error); unit: Volume per puff (ml)
Groups:
- Session 1: Own Brand Puff Volume Ad Lib: Mean ad lib puff volume: Own Brand
- Session 1: Own Brand Puff Volume Directed: Mean directed puff volume: Own Brand
- Sessions 2-5: Cowboy Vaping Liquid Puff Volume Ad Lib: Mean ad lib puff volume: Cowboy vaping liquid
- Sessions 2-5: Cowboy Vaping Liquid Puff Volume Directed: Mean directed puff volume: Cowboy vaping liquid
- Sessions 2-5: RY4 Double Vaping Liquid Puff Volume Ad Lib: Mean ad lib puff volume: RY4 Double Vaping Liquid
- Sessions 2-5: RY4 Double Vaping Liquid Puff Volume Directed: Mean directed puff volume: RY4 Double vaping liquid
- Sessions 2-5: Unflavored Vaping Liquid Puff Volume Ad Lib: Mean ad lib puff volume: Unflavored vaping liquid
- Sessions 2-5: Unflavored Vaping Liquid Puff Volume Directed: Mean directed puff volume: Unflavored vaping liquid
- Sessions 2-5: Red Oak Vaping Liquid Puff Volume Ad Lib: Mean ad lib puff volume: Red Oak vaping liquid
- Sessions 2-5: Red Oak Vaping Liquid Puff Volume Directed: Mean directed puff volume: Red Oak vaping liquid
- Session 6-7: Synthetic Nicotine Liquid Puff Volume Ad Lib: Mean ad lib puff volume: Synthetic vaping liquid
- Session 6-7: Synthetic Nicotine Liquid Puff Volume Directed: Mean directed ad lib puff volume: Synthetic vaping liquid
- Session 6-7: Tobacco Derived Liquid Puff Volume Ad Lib: Mean ad lib puff volume: Tobacco Derived vaping liquid
- Session 6-7: Tobacco Derived Liquid Puff Volume Directed: Mean directed puff volume: Tobacco Derived vaping liquid
Arm/Group | Session 1: Own Brand Puff Volume Ad Lib | Session 1: Own Brand Puff Volume Directed | Sessions 2-5: Cowboy Vaping Liquid Puff Volume Ad Lib | Sessions 2-5: Cowboy Vaping Liquid Puff Volume Directed | Sessions 2-5: RY4 Double Vaping Liquid Puff Volume Ad Lib | Sessions 2-5: RY4 Double Vaping Liquid Puff Volume Directed | Sessions 2-5: Unflavored Vaping Liquid Puff Volume Ad Lib | Sessions 2-5: Unflavored Vaping Liquid Puff Volume Directed | Sessions 2-5: Red Oak Vaping Liquid Puff Volume Ad Lib | Sessions 2-5: Red Oak Vaping Liquid Puff Volume Directed | Session 6-7: Synthetic Nicotine Liquid Puff Volume Ad Lib | Session 6-7: Synthetic Nicotine Liquid Puff Volume Directed | Session 6-7: Tobacco Derived Liquid Puff Volume Ad Lib | Session 6-7: Tobacco Derived Liquid Puff Volume Directed
Number analyzed (Participants) | 18 | 18 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17
Volume per puff (ml) | 63.5 (13.2) | 102.2 (16.1) | 66.2 (11.4) | 81.4 (14.7) | 83.6 (17.2) | 103.1 (18.6) | 63.9 (8.1) | 88.3 (13.5) | 57.5 (6.5) | 74.9 (10.61) | 86.7 (14.9) | 96.3 (13.5) | 76.9 (9.8) | 92.0 (15.2)

5. Primary Outcome: Puff Topography: Flow Rate
Description: Measure of vaping topography measuring the rate of flow per puff in milliliters per second.
Time Frame: Single Session, Approximately 2 hours in duration
Measure: Mean (Standard Error); unit: ml per second
Groups:
- Session 1: Own Brand Flow Rate Ad Lib: Mean ad lib flow rate (ml/second): Own Brand
- Session 1: Own Brand Flow Rate Directed: Mean directed flow rate (ml/second): Own Brand
- Sessions 2-5: Cowboy Vaping Liquid Flow Rate Ad Lib: Mean ad lib flow rate (ml/second): Cowboy vaping liquid
- Sessions 2-5: Cowboy Vaping Liquid Flow Rate Directed: Mean directed flow rate (ml/second): Cowboy vaping liquid
- Sessions 2-5: RY4 Double Vaping Liquid Flow Rate Ad Lib: Mean ad lib flow rate (ml/second): RY4 Double Vaping Liquid
- Sessions 2-5: RY4 Double Vaping Liquid Flow Rate Directed: Mean directed flow rate (ml/second): RY4 Double vaping liquid
- Sessions 2-5: Unflavored Vaping Liquid Flow Rate Ad Lib: Mean ad lib flow rate (ml/second): Unflavored vaping liquid
- Sessions 2-5: Unflavored Vaping Liquid Flow Rate Directed: Mean directed flow rate (ml/second): Unflavored vaping liquid
- Sessions 2-5: Red Oak Vaping Liquid Flow Rate Ad Lib: Mean ad lib flow rate (ml/second): Red Oak vaping liquid
- Sessions 2-5: Red Oak Vaping Liquid Flow Rate Directed: Mean directed flow rate (ml/second): Red Oak vaping liquid
- Session 6-7: Synthetic Nicotine Liquid Flow Rate Ad Lib: Mean ad lib flow rate (ml/second): Synthetic vaping liquid
- Session 6-7: Synthetic Nicotine Liquid Flow Rate Directed: Mean directed ad lib flow rate (ml/second): Synthetic vaping liquid
- Session 6-7: Tobacco Derived Liquid Flow Rate Ad Lib: Mean ad lib flow rate (ml/second): Tobacco Derived vaping liquid
- Session 6-7: Tobacco Derived Liquid Flow Rate Directed: Mean directed flow rate (ml/second): Tobacco Derived vaping liquid
Arm/Group | Session 1: Own Brand Flow Rate Ad Lib | Session 1: Own Brand Flow Rate Directed | Sessions 2-5: Cowboy Vaping Liquid Flow Rate Ad Lib | Sessions 2-5: Cowboy Vaping Liquid Flow Rate Directed | Sessions 2-5: RY4 Double Vaping Liquid Flow Rate Ad Lib | Sessions 2-5: RY4 Double Vaping Liquid Flow Rate Directed | Sessions 2-5: Unflavored Vaping Liquid Flow Rate Ad Lib | Sessions 2-5: Unflavored Vaping Liquid Flow Rate Directed | Sessions 2-5: Red Oak Vaping Liquid Flow Rate Ad Lib | Sessions 2-5: Red Oak Vaping Liquid Flow Rate Directed | Session 6-7: Synthetic Nicotine Liquid Flow Rate Ad Lib | Session 6-7: Synthetic Nicotine Liquid Flow Rate Directed | Session 6-7: Tobacco Derived Liquid Flow Rate Ad Lib | Session 6-7: Tobacco Derived Liquid Flow Rate Directed
Number analyzed (Participants) | 18 | 18 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17
ml per second | 28.4 (3.4) | 28.7 (3.3) | 28.2 (2.3) | 25.5 (2.7) | 29.3 (2.4) | 24.8 (2.6) | 27.8 (2.9) | 25.2 (2.8) | 27.8 (2.4) | 24.2 (1.9) | 33.7 (2.1) | 31.4 (2.1) | 33.9 (2.6) | 30.0 (2.32)

6. Secondary Outcome: Subjective Questionnaires of Product Evaluation
Description: Will be assessed by Duke Sensory Scale
Time Frame: Single Session, Approximately 2 hours in duration
Population: Mean sensory and subjective effects scores by bout type and flavor condition, Sub-Study A.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Session 1: Own Brand Ad Lib; Sessions 2-5: Cowboy Vaping Liquid Ad Lib; Sessions 2-5: RY4 Double Vaping Liquid Ad Lib; Sessions 2-5: Red Oak Vaping Liquid Ad Lib; Sessions 2-5: Unflavored Vaping Liquid Ad Lib; Sessions 6-7: Synthetic Nicotine Ad Lib; Sessions 6-7 Tobacco Derived Nicotine Liquid Ad Lib: Mean ad lib vaping topography parameters by e-liquid flavor formulation
- Session 1: Own Brand Directed; Sessions 2-5: Cowboy Vaping Liquid Directed; Sessions 2-5: RY4 Double Vaping Liquid Directed; Sessions 2-5: Red Oak Vaping Liquid Directed; Sessions 2-5: Unflavored Vaping Liquid Directed; Sessions 6-7: Synthetic Nicotine Directed; Sessions 6-7: Tobacco Derived Nicotine Liquid Directed: Mean directed vaping topography parameters by e-liquid flavor formulation
Arm/Group | Session 1: Own Brand Ad Lib | Session 1: Own Brand Directed | Sessions 2-5: Cowboy Vaping Liquid Ad Lib | Sessions 2-5: Cowboy Vaping Liquid Directed | Sessions 2-5: RY4 Double Vaping Liquid Ad Lib | Sessions 2-5: RY4 Double Vaping Liquid Directed | Sessions 2-5: Red Oak Vaping Liquid Ad Lib | Sessions 2-5: Red Oak Vaping Liquid Directed | Sessions 2-5: Unflavored Vaping Liquid Ad Lib | Sessions 2-5: Unflavored Vaping Liquid Directed | Sessions 6-7: Synthetic Nicotine Ad Lib | Sessions 6-7: Synthetic Nicotine Directed | Sessions 6-7 Tobacco Derived Nicotine Liquid Ad Lib | Sessions 6-7: Tobacco Derived Nicotine Liquid Directed
Number analyzed (Participants) | 18 | 18 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17
units on a scale
  Draw (0 "less draw" - 100 "more draw) | 72.3 (7.3) | 77.0 (5.7) | 69.7 (4.4) | 64.1 (5.6) | 61.1 (6.5) | 71.6 (4.5) | 72.9 (4.7) | 75.5 (4.2) | 68.8 (5.0) | 72.5 (4.7) | 71.9 (5.0) | 74.2 (5.3) | 66.2 (6.6) | 74.1 (5.2)
  Pleasantness (-100 "less pleasant" - +100 "more pleasant") | 45.2 (12.0) | 33.2 (15.9) | -3.2 (15.3) | -32.6 (15.5) | 3.9 (13.1) | -2.5 (13.3) | 16.4 (15.2) | 37.7 (15.7) | -2.0 (14.8) | 22.4 (16.2) | 26.2 (11.6) | 21.2 (12.9) | 1.2 (11.6) | 7.5 (14.8)
  Tingling Sensation (0 "less tingling sensation" - 100 "more tingling sensation") | 50.2 (11.4) | 34.8 (8.6) | 34.2 (6.6) | 44.4 (4.9) | 38.9 (6.5) | 44.7 (7.8) | 25.4 (5.3) | 45.1 (6.3) | 36.2 (5.6) | 33.4 (5.1) | 27.8 (5.3) | 29.8 (5.7) | 21.0 (5.2) | 29.0 (6.1)
  Product Evaluation Score: Satisfaction (1 "not at all" - 7 "extremely") | 4.8 (0.4) | 4.2 (0.4) | 2.8 (0.3) | 2.6 (0.4) | 2.7 (0.3) | 3.0 (0.4) | 3.1 (0.4) | 3.4 (0.4) | 3.1 (0.4) | 2.9 (0.4) | 3.4 (0.3) | 3.4 (0.3) | 3.1 (0.3) | 3.2 (0.3)
  Product Evaluaton Sore: Relief (1 "not at all" - 7 "extremely") | 5.3 (0.4) | 4.7 (0.6) | 3.9 (0.3) | 4.4 (0.3) | 4.0 (0.3) | 4.2 (0.3) | 4.3 (0.3) | 4.1 (0.3) | 4.5 (0.3) | 4.5 (0.3) | 4.8 (0.3) | 4.7 (0.4) | 4.4 (0.3) | 4.6 (0.3)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Session 1: Own Brand Topography Ad Lib; Session 1: Own Brand Topography Directed: SESSION 1: Participants puff their own brand liquid on study.
- Sessions 2-5: Cowboy Liquid Topography Ad Lib; Sessions 2-5: Cowboy Liquid Vaping Liquid Directed; Sessions 2-5: RY4 Vaping Liquid Topography Ad Lib; Sessions 2-5: RY4 Vaping Liquid Topography Directed; Sessions 2-5: Red Oak Vaping Liquid Topography Ad Lib; Sessions 2-5: Red Oak Vaping Liquid Topography Directed; Sessions 2-5: Unflavored Vaping Liquid Topography Ad Lib; Unflavored Vaping Liquid Vaping Topography Directed: SESSIONS 2-5: Participants puff 1 of 4 randomly assigned tobacco flavor formulations at each visit on study.
- Sessions 6-7: Synthetic Nicotine Vaping Liquid Topography Ad Lib; Sessions 6-7: Synthetic Vaping Liquid Topography Directed; Sessions 6-7: Tobacco Derived Vaping Liquid Topography Ad Lib; Sessions 6-7: Tobacco Derived Vaping Liquid Topography Directed: SESSIONS 6-7: Participants puff 1 of 2 randomly assigned nicotine formulations at each visit on study.
Arm/Group | Session 1: Own Brand Topography Ad Lib | Session 1: Own Brand Topography Directed | Sessions 2-5: Cowboy Liquid Topography Ad Lib | Sessions 2-5: Cowboy Liquid Vaping Liquid Directed | Sessions 2-5: RY4 Vaping Liquid Topography Ad Lib | Sessions 2-5: RY4 Vaping Liquid Topography Directed | Sessions 2-5: Red Oak Vaping Liquid Topography Ad Lib | Sessions 2-5: Red Oak Vaping Liquid Topography Directed | Sessions 2-5: Unflavored Vaping Liquid Topography Ad Lib | Unflavored Vaping Liquid Vaping Topography Directed | Sessions 6-7: Synthetic Nicotine Vaping Liquid Topography Ad Lib | Sessions 6-7: Synthetic Vaping Liquid Topography Directed | Sessions 6-7: Tobacco Derived Vaping Liquid Topography Ad Lib | Sessions 6-7: Tobacco Derived Vaping Liquid Topography Directed
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT05876091/Prot_SAP_001.pdf
  • Informed Consent Form (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT05876091/ICF_000.pdf